CLINICAL TRIAL: NCT00632502
Title: Safety of SCH 527123 in Subjects With Neutrophilic Asthma
Brief Title: Neutrophilic Asthma Study With Navarixin (MK-7123, SCH 527123) (MK-7123-017)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05365; 2007-005615-26 (EudraCT Number); P05365 (Other: Merck protocol number)
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Neutrophilic Asthma
MeSH Terms: interventions — navarixin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Navarixin (Experimental): Navarixin (MK-7123, SCH 527123) 30 mg capsule, to be taken by mouth once daily in the morning for 4 weeks
  Interventions: Drug: Navarixin; Drug: Rescue medication
- Placebo (Placebo Comparator): Placebo capsule to match navarixin, to be taken by mouth once daily in the morning for 4 weeks
  Interventions: Drug: Placebo; Drug: Rescue medication

INTERVENTIONS:
Drug: Navarixin — Navarixin 30 mg capsule to be taken by mouth once daily in the morning for 4 weeks.
  Arms: Navarixin
Drug: Placebo — Placebo capsule to match navarixin to be taken by mouth once daily in the morning for 4 weeks.
  Arms: Placebo
Drug: Rescue medication — Participant choice of short-acting beta-2 agonist (salbutamol/albuterol), anticholinergic, or combination medication as needed for asthma symptoms

SUMMARY:
4-Week Safety Study in Subjects with Neutrophilic Asthma

DETAILED DESCRIPTION:
Effect of treatment with navarixin (MK-7123, SCH 527123) on sputum neutrophils and asthma symptoms

ELIGIBILITY:
Inclusion Criteria:

* 18 to <=70 years of age, either sex, any race.
* Induced sputum neutrophil count >=40% of total white blood cells and <10 million/mL at Screening.
* Documented diagnosis of asthma (within past 5 years), determined by at least one of the following: >=12% and 200 mL improvement in Forced Expiratory Volume in 1 second (FEV1) post-bronchodilator, and/or airway hyperresponsiveness (eg, positive methacholine challenge <8 mg/mL).
* Nonsmoker or previous smoker with cumulative smoking history less than 20 pack-years (pack-year = 20 cigarettes smoked daily for 1 year). Previous smokers may not have smoked within 1 year prior to Screening.
* Must not have had an exacerbation of asthma for 4 weeks prior to Screening and must be on a stable medication regimen for asthma at least 4 weeks prior to Screening.
* Must be receiving >=800 mcg/day of beclomethasone dipropionate (BDP) or equivalent for at least 3 months prior to Screening (and on stable dose for at least 4 weeks prior to Screening).
* Must be willing to give written informed consent to participate in the study
* Must be capable of complying with the dosing regimen, adhere to the visit schedule, and participate in all treatment procedures, including sputum induction.
* Female subject of childbearing potential must have a negative serum pregnancy test at Screening and must be using a medically acceptable, highly effective, adequate form of birth control (ie, failure rate <1% per year when used consistently and correctly) prior to Screening and agree to continue using it while in the study (Screening and Treatment Periods). Medically acceptable, highly effective forms of birth control are hormonal implants, oral contraceptives, medically acceptable prescribed intrauterine devices (IUDs), and monogamous relationship with a male partner who has had a vasectomy. Female subject who is not of childbearing potential must have a medical record of being surgically sterile (eg, hysterectomy, tubal ligation), or be at least 1 year postmenopausal. Absence of menses for at least 1 year will indicate that a female is postmenopausal. A female subject should be encouraged to continue using a highly effective method of birth control for 30 days following the end of treatment.
* Male subject must agree to use an adequate form of contraception for the duration of the study and agree to have sexual relations only with women who use a highly effective birth control method.

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD)/other relevant lung disease (other than asthma).
* 4 weeks prior to/or Screening: upper/lower respiratory tract infection.
* Prohibited medications received more recently than indicated washout prior to Screening
* Screening: Inadequate amount or difficulty producing sputum.
* Screening: Sputum neutrophil count over 10 million/mL.
* Screening: peripheral blood neutrophil (PBN) count <3000/µL.
* Post-bronchodilator FEV1 <1L.
* Clinically significant chronic infectious disease(s) (eg, Human Immunodeficiency Virus [HIV], hepatitis B or C).
* Allergy/sensitivity to study drug/excipients.
* Breast-feeding, pregnant/intends to become pregnant during study.
* Requiring mechanical ventilation for respiratory event within 6 months of Screening.
* Medical condition(s) (eg, hematologic, cardiovascular, renal, hepatic, neurologic, or metabolic) or medication that may interfere with effect of study medication.
* Within 30 days of Screening: any other investigational drug.
* Participation in any other clinical study.
* Part of the staff personnel involved with the study.
* Family member of investigational study staff.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2009-02-01 (Actual); Study Completion 2009-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Nair P, Gaga M, Zervas E, Alagha K, Hargreave FE, O'Byrne PM, Stryszak P, Gann L, Sadeh J, Chanez P; Study Investigators. Safety and efficacy of a CXCR2 antagonist in patients with severe asthma and sputum neutrophils: a randomized, placebo-controlled clinical trial. Clin Exp Allergy. 2012 Jul;42(7):1097-103. doi: 10.1111/j.1365-2222.2012.04014.x. PMID 22702508
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P05365&kw=7123-017&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered to complete the study if they completed the follow-up visit, whether or not they completed treatment.
Groups:
- Navarixin: Navarixin 30 mg capsule to be taken by mouth once daily for 4 weeks
- Placebo: Placebo capsule to be taken by mouth once daily for 4 weeks
Period: Overall Study
Arm/Group | Navarixin | Placebo
Started | 25 | 12
Treated | 22 | 12
Completed Treatment | 19 | 9
Completed | 22 | 11
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Randomized not treated | 3 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Navarixin | Placebo | Total
Number analyzed (Participants) | 22 | 12 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.7 (10.6) | 53.9 (6.8) | 50.6 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Maintained an Absolute Peripheral Blood Neutrophil Count >=1500/µL
Description: Peripheral blood neutrophil counts were performed on Day 2 and Weeks 1, 2, 3, and 4 of the treatment period
Time Frame: Up to 4 weeks
Population: The analysis population included all participants who received at least one dose of study drug
Measure: Number; unit: Number of participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 22 | 12
Number of participants | 20 | 12

2. Secondary Outcome: Mean Change From Baseline in Sputum Absolute Neutrophil Count
Description: Induced sputum samples were obtained at Baseline and at Weeks 2 and 4 of the treatment period. Samples were collected before study drug administration using the nebulizer method and sent to a central laboratory for analysis. An average was taken over all post-baseline samples collected no later than one day after the last dose of study drug.
Time Frame: Baseline and while on study drug (up to 4 weeks)
Population: The analysis population included all randomized participants who received at least one dose of study drug and had sputum absolute neutrophil counts at Baseline or Week 4
Measure: Mean (Standard Deviation); unit: Neutrophil count X10^9/L
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 18 | 11
Neutrophil count X10^9/L
  Baseline sputum absolute neutrophil count | 3.275 (3.995) | 3.408 (2.973)
  Change from baseline at up to 4 weeks | -0.270 (6.673) | 0.680 (2.249)

3. Secondary Outcome: Mean Change From Baseline in Total Asthma Symptom Score
Description: Total Asthma Symptom Score is the sum of individual symptoms of wheezing, coughing, and dyspnea assessed twice daily (morning and evening) and is recorded on a comment diary card. Each of the symptoms receives a daily score from 0 (none) to 3 (severe), averaged over the two daily assessments. The total score ranges from 0 to 9, with a lower score indicating less severe asthma symptoms.
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: The analysis population included all randomized participants who received at least one dose of study drug and had Asthma Symptom Scores evaluated at the time points reported
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Navarixin: Navarixin (SCH 537123) 30 mg capsule to be taken by mouth once daily for 4 weeks
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 21 | 12
Score on a scale
  Baseline Total Asthma Symptom Score (n=21, 12) | 2.47 (1.83) | 2.40 (1.30)
  Change at 1 week (n=21, 12) | -0.07 (1.01) | 0.05 (0.78)
  Change at 2 weeks (n=20, 12) | -0.25 (1.50) | 0.19 (1.14)
  Change at 3 weeks (n=19, 12) | -0.19 (1.56) | 0.04 (1.30)
  Change at 4 weeks (n=18, 9) | -0.00 (1.62) | -0.26 (2.06)

4. Secondary Outcome: Change From Baseline in Post-Bronchodilator Forced Expiratory Volume in One Second (FEV1)
Description: Spirometry was used to measure post-bronchodilator FEV1 at Baseline and before study drug administration at Weeks 1, 2, 3, and 4. Participants received 4 puffs of bronchodilator (salbutamol hydrofluoroalkane or equivalent) at 30-second intervals and spirometry was performed 30 minutes later. The mean change from baseline is based on the average change over all post-baseline assessments.
Time Frame: Baseline and up to 4 weeks
Population: The analysis population included all randomized participants who received at least one dose of study drug and had endpoint assessment at Baseline or at any post-baseline visit
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 22 | 12
Liters
  Baseline FEV1 | 2.197 (0.948) | 1.851 (0.469)
  Average change from baseline at up to 4 weeks | -0.099 (0.315) | -0.094 (0.106)

5. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire With Standardized Activities (AQLQ[S])
Description: The AQLQ[S] was administered at Baseline and at Weeks 2 and 4. The assessment consists of a 32-item questionnaire covering 4 domains: symptoms, emotional functioning, impact of environmental stimuli, and activity limitation. Each item receives a score from 1 (worst, or most affected) to 7 (not at all affected). The score is the mean across all items, and ranges from 1 to 7. The mean change from baseline is based on the average change over all post-baseline assessments.
Time Frame: Baseline and up to 4 weeks
Population: The analysis population included all randomized participants who received at least one dose of study drug and had endpoint evaluation at Baseline or at any post-baseline visit
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 21 | 12
Score on a scale
  Baseline AQLQ[S] Score | 4.822 (1.568) | 4.897 (1.128)
  Average change from baseline at up to 4 weeks | 0.165 (0.901) | 0.119 (0.936)

6. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Up to 5 weeks
Population: The analysis population included all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 22 | 12
Participants | 13 | 8

7. Secondary Outcome: Number of Participants With an Electrocardiogram Adverse Event
Description: The endpoint measured was any electrocardiogram abnormality that was reported as an AE. An AE is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Week 4
Population: The analysis population included all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 22 | 12
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With a Laboratory Adverse Event
Description: The endpoint measured was any laboratory (hematology, blood chemistry, or urinalysis) abnormality that was reported as an AE. An AE is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions.
Time Frame: Up to 5 weeks
Population: The analysis population included all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 22 | 12
Participants | 2 | 0

9. Secondary Outcome: Number of Participants Who Discontinued the Study Because of an Adverse Event
Description: as for outcome 6
Time Frame: Up to 5 weeks
Population: The analysis population included all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 22 | 12
Participants | 0 | 1

10. Secondary Outcome: Number of Participants Who Discontinued Treatment Because of an Adverse Event or a Protocol-defined Clinical Event
Description: An AE is any untoward medical occurrence in a participant administered study drug which does not necessarily have a causal relationship with the treatment. AEs may include the onset of new illness and the exacerbation of pre-existing conditions. A protocol-defined clinical event is an asthma exacerbation requiring addition of or increase in systemic steroids, as determined by the investigator.
Time Frame: Up to 4 weeks
Population: The analysis population included all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 22 | 12
Participants
  Adverse event | 2 | 2
  Protocol-defined clinical event | 1 | 1

11. Secondary Outcome: Maximum Plasma Concentration of Navarixin (Cmax)
Description: Plasma samples were to be collected at baseline and up to 24 hours after dosing with navarixin at Weeks 1, 2, 3, and 4
Time Frame: Week 1, 2, 3, and 4
Population: The analysis population was to include all participants who received at least one dose of navarixin and had navarixin plasma concentrations available for endpoint evaluation. The planned outcome measure was not evaluated.
Arm/Group | Navarixin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 weeks
Arm/Group | Navarixin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 11/22 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin (N=22) | Placebo (N=12)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.